CLINICAL TRIAL: NCT07386535
Title: Innovative Tools to Expand Music-Inspired Strategies for Blood Pressure and Stroke Prevention
Acronym: ITEST-BPStroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Nigerian Institute of Medical Research (Other Government); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 202403128; R01HL168766 (NIH)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: High Blood Pressure; Stroke
Keywords: High blood pressure; Stroke; Hypertension; Young people; Adult caregivers; Prevention
MeSH Terms: conditions — Hypertension; Stroke

STUDY DESIGN:
Intervention Model Description: Hybrid Type II stepped-wedge cluster randomized trial
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music4Health Intervention (Experimental): Each of the 30 local government areas (LGAs) will be randomly allocated using block randomization to one of the four waves, with 7-8 LGAs allocated to each wave. All waves will begin with a control period with the first wave commencing the intervention period three months following the study start and each subsequent wave commencing one month following the start date of the previous wave's intervention period. Each wave's intervention period will last three months.
  Interventions: Behavioral: Music4Health Intervention

INTERVENTIONS:
Behavioral: Music4Health Intervention — The intervention period will include three Music4Health Day community events. Music4Health Day will adapt content from open call submissions and apprenticeships with community-based teams to meet the music preferences of youth and their caregivers. The events will focus on managing blood pressure, preventing strokes, and stroke preparedness through music-inspired strategies, utilizing rhythms and lyrics. Each Music4Health Day event will include a listening session of a music video with lyrics designed to improve knowledge and awareness of high blood pressure and stroke preparedness. Participants will be provided with MP3 files and YouTube video links containing music, videos, visuals, and health messages. Participants will listen to the intervention at the events and also at their convenience on their mobile phones, followed by weekly text reminders. During the events, music ambassadors will also share personal experiences to promote health messages and foster community engagement.
  Other Names: Implementation Phase

SUMMARY:
Expanding evidence-based interventions for hypertension and stroke prevention among youth and their caregivers is crucial for meeting World Health Organization and Nigerian health goals. Innovative strategies are urgently needed to address the burden of hypertension and stroke in Nigeria, aiming to involve local communities, bridge generational gaps, and reduce health disparities. This study aims to determine the effect of a music-inspired intervention and campaign (Music4Health) designed by the community on blood pressure, stroke preparedness and intentions, and uptake of the intervention among youth-caregiver dyads in Nigeria.

DETAILED DESCRIPTION:
This study will be a stepped-wedge cluster randomized controlled trial conducted in 30 local government areas in Nigeria. The aim of the study will be to test if the music-inspired intervention reduces blood pressure in caregivers ≥40 years old, maintains blood pressure in youth 14-24 years old, and improves stroke preparedness among youth and caregivers. Sites will be randomly assigned to one of four waves, which will deliver the intervention to a longitudinal cohort of youth-caregiver dyads, spaced one month between each wave. The control period will last three months and include no intervention, and the intervention period will last three months for each wave and will include three music listening sessions (Music4Health Day) spaced one month apart. Participants will be recruited and enrolled in the trial through various methods, including community outreach, referrals, and social media. Participants will be invited to attend three community-based Music4Health Days on predetermined dates (schedule based on randomized intervention waves) and will be asked to return to the intervention site for follow-up data collection, including blood pressure measurements and validated questionnaires. The Music4Health Day intervention will include a listening session of a music video with lyrics designed to improve knowledge and awareness of high blood pressure and stroke preparedness. During Music4Health Day, music ambassadors will also share personal experiences to promote health messages and foster community engagement. Following the intervention period, the investigators will follow the cohort for six months after the intervention period to collect outcome data from each participant.

ELIGIBILITY:
Inclusion Criteria:

Youth Participants

* Aged 14-24 years
* Reside in one of the 30 selected LGAs
* Able to provide informed consent
* Willing to participate in the M4H campaign

Caregiver Participants

* Aged ≥40 years
* Identified as a caregiver (biological/surrogate parent, grandparent, or close relative)
* Reside in the same household or have a caregiving relationship with eligible youth
* Able to provide informed consent

General Eligibility for Dyads

* Must be a youth-caregiver dyad (one youth and one caregiver)
* Both members must consent to participate and complete baseline assessments
* Reside in or be affiliated with the selected study LGAs

Exclusion Criteria:

Youth Participants

* Below 14 or above 24 years
* Inability to provide informed consent
* Unwilling to participate in intervention activities

Caregiver Participants

* Below 40 years of age
* Not serving in a caregiver role to eligible youth
* Inability to provide informed consent

General Eligibility for Dyads

* Either party of the dyad does not meet the inclusion criteria
* Refusal to participate or complete baseline assessments

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1412 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2027-10-26 (Estimated); Study Completion 2027-10-26 (Estimated)

PRIMARY OUTCOMES:
Maintenance of normal blood pressure for youth participants | Months 0, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14
  Systolic and diastolic blood pressure will be collected by trained research facilitators. A normal blood pressure among youth is defined as <120/80 mmHg.
Systolic blood pressure reduction for caregiver participants | Months 0, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14
  Systolic and diastolic blood pressure will be collected by trained research facilitators.
Stroke preparedness knowledge for youth and caregiver participants | Months 0, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14
  Stroke preparedness knowledge is defined as the ability to recognize signs of stroke (i.e., F.A.S.T. warning signs) and the intention to seek treatment immediately. Their knowledge will be ascertained by self-report using surveys.
Uptake of music-inspired hypertension/stroke prevention campaign (Music4Health) among youth and caregiver participants | Months 0, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14
  Uptake of the campaign is defined as the absolute number, proportion, and representativeness of participants who participate in the campaign (i.e., attend listening sessions).

SECONDARY OUTCOMES:
Intervention Acceptability | Months 0, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14
  This will measure the ITEST BP/Stroke campaign. Measured using the Acceptability of Intervention Measure (AIM), Cronbach's alpha = 0.85. The four item measure participants' satisfaction, important implementation outcomes that are often considered a "leading indicator" of implementation success. The subscales are rated on a 5-point Likert scale, 1 to 5, with higher scores indicating higher acceptability. This will be measured using a self-administered questionnaire and in-depth interviews facilitated by trained research staff.
Intervention Fidelity | Months 0, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14
  This will measure the evidence that the core ITEST BP/Stroke campaign components were delivered as intended in relation to the study protocol, consistency of implementation across 30 study sites (LGAS). This will be assessed both quantitatively and qualitatively using the following four dimensions: (1) Frequency: number of intervention-related interactions; (2) Duration: length of each component of the intervention; (3) Content: the knowledge or behavioral change the music-inspired intervention seeks to deliver to the youth and caregiver dyads; and (4) Coverage: the number of youth/caregiver dyads who receive the music-inspired intervention as intended over the number of participants who are enrolled. This will be measured using a self-administered questionnaire and in-depth interviews facilitated by trained research staff.
Intervention Reach | Months 0, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14
  The proportion of eligible youth/caregiver dyads reached versus the total target population. Measured as 1) the participation rate among eligible participants; 2) the representativeness of participants based on demographic and health characteristics. The reasons given for declining to participate will also be assessed. This will be measured using a self-administered questionnaire and in-depth interviews facilitated by trained research staff.
Intervention Sustainment | Months 0, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14
  This will measure the maintenance of the BP/Stroke campaign using the Stages of Implementation Completion (SIC), an eight-stage assessment tool will be used to assess the sustainment of the intervention. This tool delineates the start of implementation. This will be measured using a self-administered questionnaire and in-depth interviews facilitated by trained research staff.

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Iwelunmor, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Nigerian Institute of Medical Research, Yaba, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trappe HJ. The effects of music on the cardiovascular system and cardiovascular health. Heart. 2010 Dec;96(23):1868-71. doi: 10.1136/hrt.2010.209858. PMID 21062776
- [Background] Braveman P, Egerter S, Williams DR. The social determinants of health: coming of age. Annu Rev Public Health. 2011;32:381-98. doi: 10.1146/annurev-publhealth-031210-101218. PMID 21091195
- [Background] Bigna JJ, Noubiap JJ. The rising burden of non-communicable diseases in sub-Saharan Africa. Lancet Glob Health. 2019 Oct;7(10):e1295-e1296. doi: 10.1016/S2214-109X(19)30370-5. No abstract available. PMID 31537347
- [Background] Ajayi S, Adebiyi A, Kadiri S. Increased urinary sodium excretion is associated with systolic blood pressure in first degree relatives of hypertensive patients in Ibadan, Southwestern Nigeria. Pan Afr Med J. 2018 Nov 9;31:168. doi: 10.11604/pamj.2018.31.168.16611. eCollection 2018. PMID 31086621
- [Background] Akinyemi RO, Ovbiagele B, Adeniji OA, et al. Stroke in Africa: profile, progress, prospects and priorities. Nature Reviews Neurology. 2021;17(10):634-656.
- [Background] Sarfo FS, Ovbiagele B, Gebregziabher M, et al. Stroke among young West Africans: evidence from the SIREN (Stroke Investigative Research and Educational Network) large multisite case-control study. Stroke. 2018;49(5):1116-1122.